CLINICAL TRIAL: NCT04650776
Title: Single-centre Experimental Evaluation of Methods for Reliable Non-invasive Prediction of Thermal Strain in Healthy Male Adults
Brief Title: Non-invasive Prediction of Thermal Strain in Healthy Male Adults
Acronym: HUMONHEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Annaheim (Other)
Responsible Party: Sponsor-Investigator, Simon Annaheim, Principal Investigator, Empa, Swiss Federal Laboratories for Materials Science and Technology
Organization: Empa, Swiss Federal Laboratories for Materials Science and Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 5213.00095
Record Dates: First submitted 2020-11-19; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Heat Stress
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High heat strain (Experimental): participants exercised at 75% of their heart rate maximum (HR max) and wore light athletic clothing (t-shirt and shorts)
  Interventions: Other: Heat strain
- Low heat strain (Experimental): participants exercised at 50% HR max, wearing protective firefighter clothing (jacket and trousers)
  Interventions: Other: Heat strain

INTERVENTIONS:
Other: Heat strain — The experimental procedure comprised 15 min baseline seated rest (23.2 ± 0.3°C, 24.5 ± 1.6% relative humidity), followed by 15 min seated rest and cycling in a climatic chamber (35.4 ± 0.2◦C, 56.5 ± 3.9% relative humidity; to +1.5◦C or maximally 38.5°C rectal temperature, duration 20-60 min), with a final 30 min seated rest outside the chamber.

SUMMARY:
This is primarily an experimental study investigating methods of temperature measurement / heat strain detection. In the calibration study, there are different skin temperature sensor types, and in the prediction study there are different methods for determining heat strain, including conventional methods (rectal, gastro-intestinal), the development of a prediction model, and an index based on heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy males
* aged 18-45 y
* regularly participate in sport, exercise, or equivalent physical activity on a weekly basis.

Exclusion Criteria:

* Known injuries or illnesses that may affect safe participation. These include injuries or illnesses involving (but not limited to):
* cardiovascular, renal, or gastrointestinal tract
* heat or exercise intolerance
* acute infections,
* immunological diseases (including asthma)
* psychiatric disorders.
* Participants must not be currently or previously on cardiovascular-related medication and must not be taking psychotropic medication (last 60 days).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Core body temperature | 90 minutes
  Rectal core body temperature (unit of measure is degree celsius °C)
Predicted core body temperature | 90 minutes
  Estimated core body temperature (°C) from selected non-invasive measurements: applying a multiple linear regression model several predictive parameters, including skin temperature at different body sites, heat flux at different body sites, and heart rate will be combined to achieve one reported temperature value (°C)
ECG-based heat strain index | 90 minutes
  ECG-based index of heat strain derived from heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Simon Annaheim, Dr., Principal Investigator — Empa, Swiss Federal Laboratories for Materials Science and Technology
Locations (1):
- Empa, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data is available upon request from qualified researchers.

REFERENCES:
- See also: Published manuscript — https://www.frontiersin.org/articles/10.3389/fphys.2018.01780/full